CLINICAL TRIAL: NCT05664607
Title: The Impact of Sarcopenia and the Effect of Multimodal Rehabilitation on the Prognosis of Rectal Cancer Patients Receiving Concurrent Chemoradiotherapy- Randomized Controlled Trial
Brief Title: Sarcopenia and Multimodal Rehabilitation on the Prognosis of Rectal Cancer Patients Receiving CCRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wan-Hsiang Hu, Attending physician, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202200748A3
Record Dates: First submitted 2022-11-29; First posted 2022-12-23 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; concurrent chemoradiotherapy; sarcopenia; multimodal rehabilitation
MeSH Terms: conditions — Rectal Neoplasms; Sarcopenia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): no multimodal rehabilitation
- multimodal rehabilitation group (Experimental): include excise, nutrition consultant, nutrition supplement and psychologic intervention.
  Interventions: Other: for excise, nutrition consultant, nutrition supplement and psychologic intervention.

INTERVENTIONS:
Other: for excise, nutrition consultant, nutrition supplement and psychologic intervention. — for excise, nutrition consultant, nutrition supplement and psychologic intervention.
  Arms: multimodal rehabilitation group

SUMMARY:
Investigators use clinical trial to explore the role of sarcopenia and multimodal rehabilitation in prognosis of rectal cancer patients receiving concurrent chemoradiotherapy.

DETAILED DESCRIPTION:
The impact of sarcopenia and the effect of multimodal rehabilitation will be evaluated in the rectal cancer patients receiving pre-operative concurrent chemoradiotherapy. This is a randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* age>20
* rectal cancer patients receiving concurrent chemoradiotherapy
* agree to join the trial and sign the informed consent form

Exclusion Criteria:

* unstable vital sign
* unable to excise
* not suitable after evaluation by Principal Investigator

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Sarcopenia assessment with muscle power | baseline
  Assessment with Grip strength(Kg)
Sarcopenia assessment with muscle power | 1.5 months later
  Assessment with Grip strength(Kg)
Sarcopenia assessment with muscle power | 3 months later
  Assessment with Grip strength(Kg)
Sarcopenia assessment with speed | baseline
  Assessment with speed(m/s)
Sarcopenia assessment with speed | 1.5 months later
  Assessment with speed(m/s)
Sarcopenia assessment with speed | 3 months later
  Assessment with speed(m/s)
Sarcopenia assessment with DXA | baseline
  Assessment with DXA(g/cm2)
Sarcopenia assessment with DXA | 3 months later
  Assessment with DXA(g/cm2)
Sarcopenia assessment with abdominal CT | baseline
  Assessment with ASM/heigh2(Kg/m2) of L3 level
Sarcopenia assessment with abdominal CT | 3 months later
  Assessment with ASM/heigh2(Kg/m2) of L3 level
Nutrition assessment with albuminemia | baseline
  albumin level in serum
Nutrition assessment with albuminemia | 1.5 months later
  albumin level in serum
Nutrition assessment with albuminemia | 3 months later
  albumin level in serum
Nutrition assessment with pre-albuminemia | baseline
  pre-albumin level in serum
Nutrition assessment with pre-albuminemia | 1.5 months later
  pre-albumin level in serum
Nutrition assessment with pre-albuminemia | 3 months later
  pre-albumin level in serum
Nutrition assessment with PGSGA | baseline
  patient-generated subjective global assessment Scale (Total score 0~9
  ;score 1-3 Good nutritional intake. score 4-8 Moderate malnutrition. score >9Severe malnutrition)
Nutrition assessment with PGSGA | 1.5 months later
  patient-generated subjective global assessment Scale (Total score 0~9
  ;score 1-3 Good nutritional intake. score 4-8 Moderate malnutrition. score >9Severe malnutrition)
Nutrition assessment with PGSGA | 3 months later
  patient-generated subjective global assessment Scale (Total score 0~9
  ;score 1-3 Good nutritional intake. score 4-8 Moderate malnutrition. score >9Severe malnutrition)
Psychological assessment | baseline
  Taiwanese Depression Questionnaire (TDQ)Total score 0-54; score >8 emotionally stable ;Score 9 ~ 14 Pay attention to emotional changes Score 15 ~ 18 pressure load reaches the critical point; Score 19-28 It is recommended to find a professional institution or medical unit assistance
  ;Scores 29 or more must find professional medical units to get involved
Psychological assessment | 1.5 months later
  Taiwanese Depression Questionnaire (TDQ)Total score 0-54; score >8 emotionally stable ;Score 9 ~ 14 Pay attention to emotional changes Score 15 ~ 18 pressure load reaches the critical point; Score 19-28 It is recommended to find a professional institution or medical unit assistance
  ;Scores 29 or more must find professional medical units to get involved
Psychological assessment | 3 months later
  Taiwanese Depression Questionnaire (TDQ)Total score 0-54; score >8 emotionally stable ;Score 9 ~ 14 Pay attention to emotional changes Score 15 ~ 18 pressure load reaches the critical point; Score 19-28 It is recommended to find a professional institution or medical unit assistance
  ;Scores 29 or more must find professional medical units to get involved
Harris Benedict Equation | baseline
  Total Daily Energy Expenditure
Harris Benedict Equation | 1.5 months later
  Total Daily Energy Expenditure
Harris Benedict Equation | 3 months later
  Total Daily Energy Expenditure

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Hsiang Hu, Principal Investigator — Chang Gung Memorial Hospital,Kaohsiung, Taiwan, 833
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Lieffers JR, Bathe OF, Fassbender K, Winget M, Baracos VE. Sarcopenia is associated with postoperative infection and delayed recovery from colorectal cancer resection surgery. Br J Cancer. 2012 Sep 4;107(6):931-6. doi: 10.1038/bjc.2012.350. Epub 2012 Aug 7. PMID 22871883
- [Background] Reisinger KW, van Vugt JL, Tegels JJ, Snijders C, Hulsewe KW, Hoofwijk AG, Stoot JH, Von Meyenfeldt MF, Beets GL, Derikx JP, Poeze M. Functional compromise reflected by sarcopenia, frailty, and nutritional depletion predicts adverse postoperative outcome after colorectal cancer surgery. Ann Surg. 2015 Feb;261(2):345-52. doi: 10.1097/SLA.0000000000000628. PMID 24651133
- [Background] Choi MH, Oh SN, Lee IK, Oh ST, Won DD. Sarcopenia is negatively associated with long-term outcomes in locally advanced rectal cancer. J Cachexia Sarcopenia Muscle. 2018 Feb;9(1):53-59. doi: 10.1002/jcsm.12234. Epub 2017 Aug 28. PMID 28849630
- [Background] Nakanishi R, Oki E, Sasaki S, Hirose K, Jogo T, Edahiro K, Korehisa S, Taniguchi D, Kudo K, Kurashige J, Sugiyama M, Nakashima Y, Ohgaki K, Saeki H, Maehara Y. Sarcopenia is an independent predictor of complications after colorectal cancer surgery. Surg Today. 2018 Feb;48(2):151-157. doi: 10.1007/s00595-017-1564-0. Epub 2017 Jul 11. PMID 28699003
- [Background] Chen LK, Liu LK, Woo J, Assantachai P, Auyeung TW, Bahyah KS, Chou MY, Chen LY, Hsu PS, Krairit O, Lee JS, Lee WJ, Lee Y, Liang CK, Limpawattana P, Lin CS, Peng LN, Satake S, Suzuki T, Won CW, Wu CH, Wu SN, Zhang T, Zeng P, Akishita M, Arai H. Sarcopenia in Asia: consensus report of the Asian Working Group for Sarcopenia. J Am Med Dir Assoc. 2014 Feb;15(2):95-101. doi: 10.1016/j.jamda.2013.11.025. PMID 24461239
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Bano G, Trevisan C, Carraro S, Solmi M, Luchini C, Stubbs B, Manzato E, Sergi G, Veronese N. Inflammation and sarcopenia: A systematic review and meta-analysis. Maturitas. 2017 Feb;96:10-15. doi: 10.1016/j.maturitas.2016.11.006. Epub 2016 Nov 13. PMID 28041587
- [Background] Lin JX, Lin JP, Xie JW, Wang JB, Lu J, Chen QY, Cao LL, Lin M, Tu R, Zheng CH, Huang CM, Li P. Prognostic Value and Association of Sarcopenia and Systemic Inflammation for Patients with Gastric Cancer Following Radical Gastrectomy. Oncologist. 2019 Nov;24(11):e1091-e1101. doi: 10.1634/theoncologist.2018-0651. Epub 2019 Mar 25. PMID 30910865
- [Background] Tessier AJ, Chevalier S. An Update on Protein, Leucine, Omega-3 Fatty Acids, and Vitamin D in the Prevention and Treatment of Sarcopenia and Functional Decline. Nutrients. 2018 Aug 16;10(8):1099. doi: 10.3390/nu10081099. PMID 30115829
- [Background] Minnella EM, Bousquet-Dion G, Awasthi R, Scheede-Bergdahl C, Carli F. Multimodal prehabilitation improves functional capacity before and after colorectal surgery for cancer: a five-year research experience. Acta Oncol. 2017 Feb;56(2):295-300. doi: 10.1080/0284186X.2016.1268268. Epub 2017 Jan 12. PMID 28079430
- [Background] Gillis C, Li C, Lee L, Awasthi R, Augustin B, Gamsa A, Liberman AS, Stein B, Charlebois P, Feldman LS, Carli F. Prehabilitation versus rehabilitation: a randomized control trial in patients undergoing colorectal resection for cancer. Anesthesiology. 2014 Nov;121(5):937-47. doi: 10.1097/ALN.0000000000000393. PMID 25076007
- [Background] Barberan-Garcia A, Ubre M, Roca J, Lacy AM, Burgos F, Risco R, Momblan D, Balust J, Blanco I, Martinez-Palli G. Personalised Prehabilitation in High-risk Patients Undergoing Elective Major Abdominal Surgery: A Randomized Blinded Controlled Trial. Ann Surg. 2018 Jan;267(1):50-56. doi: 10.1097/SLA.0000000000002293. PMID 28489682
- [Background] Hu WH, Chang CD, Liu TT, Chen HH, Hsiao CC, Kang HY, Chuang JH. Association of sarcopenia and expression of interleukin-23 in colorectal cancer survival. Clin Nutr. 2021 Oct;40(10):5322-5326. doi: 10.1016/j.clnu.2021.08.016. Epub 2021 Aug 30. PMID 34536640